CLINICAL TRIAL: NCT04996940
Title: Comparative Acceptability of Tobacco and Menthol Flavored E-cigarettes Among Menthol Cigarette Smokers
Brief Title: Comparative Acceptability of Tobacco and Menthol Flavored E-cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 145421a
Record Dates: First submitted 2021-07-14; First posted 2021-08-09 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Tobacco Use Disorder
Keywords: tobacco; e-cigarette
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Intervention Model Description: Participants will then be randomized 1:1 to e-cigarette flavor order (tobacco e-cigarette, menthol e-cigarette). They will complete a 30-minute ad libitum session with the first product, based on randomization, followed by a 1.5 hour standard washout period, followed by a 30-minute ad libitum vaping session with the second product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tobacco then Menthol (Experimental): A 30-minute session with tobacco flavor then a 30-min session with menthol flavor
  Interventions: Device: E-cigarette product
- Menthol then tobacco (Experimental): A 30-minute session with menthol flavor then a 30-min session with tobacco flavor
  Interventions: Device: E-cigarette product

INTERVENTIONS:
Device: E-cigarette product — Participants will be randomized 1:1 to e-cigarette flavor order either:
  1. tobacco e-cigarette
  2. menthol e-cigarette

SUMMARY:
The study is a randomized crossover trial. Current menthol smokers will complete a session with each flavor of an electronic cigarette: menthol and tobacco. The objective of this survey is to assess for flavor preference.

DETAILED DESCRIPTION:
Participants who report typically smoking menthol cigarettes will be invited to complete a session. Participants will undergo overnight tobacco/nicotine abstinence before the visit (eCO<12ppm). Participants will then be randomized 1:1 to e-cigarette flavor order (tobacco e-cigarette, menthol e-cigarette). They will complete a 30-minute ad libitum session with the first product, based on randomization, followed by a 1.5 hour standard washout period, followed by a 30-minute ad libitum vaping session with the second product. Throughout each session, puff topography will be measured via a pressure sensor attached to the e-cigarette device. Participants will complete self-report measures of smoking urges and withdrawal symptoms pre- and post-vaping session. In addition, they will complete measures of subjective vaping experience, perceptions of flavor, product demand, and intentions for future use.

ELIGIBILITY:
Inclusion Criteria:

* typically smoking menthol cigarettes
* Non-Hispanic African American or white/Caucasian,
* ≥21 years old, smoke 5-30 cigarettes per day,
* daily cigarette smoker
* smoked at current rate for at least 6 months
* interested in trying e-cigarettes
* not interested in or unable/unwilling to quit cigarette smoking
* willing to complete one in-person study visits

Exclusion Criteria:

* Interested in quitting cigarettes in the next 30 days
* use of smoking cessation pharmacotherapy in the past 30 days
* use of non-cigarette tobacco products in the past 30 days
* use of e-cigarettes >5x in lifetime
* use of e-cigarettes ≥4 of the past 30 days
* weight < 110 lbs
* uncontrolled hypertension (systolic BP ≥ 180 or diastolic BP ≥ 105)
* pregnant, plans to become pregnant, or breastfeeding
* live >10 miles from study site (Fairway CRU)
* current enrollment is a research study or program that aims to alter tobacco use

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tobacco Flavor Pod Then Menthol Flavor Pod: At lab visit 1 participant receive tobacco flavored pod for the electronic cigarette during the during the 30 minute session with the electronic cigarette. The researcher and participant were blinded to flavor during the visit.
  Following at least a 48-hour washout period, at lab visit 2, receive menthol flavored pod for the electronic cigarette during the 30 minute session with the electronic cigarette. The researcher and participant were blinded to flavor during the visit.
- Menthol Flavor Pod Then Tobacco Flavor Pod: At lab visit 1 participant receive menthol flavored pod for the electronic cigarette during the 30 minute session with the electronic cigarette. The researcher and participant were blinded to flavor during the visit.
  Following at least a 48-hour washout period, at lab visit 2, receive tobacco flavored pod for the electronic cigarette during the 30 minute session with the electronic cigarette. The researcher and participant were blinded to flavor during the visit.
Period: Overall Study
Arm/Group | Tobacco Flavor Pod Then Menthol Flavor Pod | Menthol Flavor Pod Then Tobacco Flavor Pod
Started | 28 | 24
Completed | 28 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tobacco Then Menthol: A 30-minute session with tobacco flavor then a 30-min session with menthol flavor
  E-cigarette product: Participants will be randomized 1:1 to e-cigarette flavor order either:
  1. tobacco e-cigarette
  2. menthol e-cigarette
- Menthol Then Tobacco: A 30-minute session with menthol flavor then a 30-min session with tobacco flavor
  E-cigarette product: Participants will be randomized 1:1 to e-cigarette flavor order either:
  1. tobacco e-cigarette
  2. menthol e-cigarette
- Total: Total of all reporting groups
Arm/Group | Tobacco Then Menthol | Menthol Then Tobacco | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Continuous [Mean (Full Range); unit: years] | 54.0 [32 to 70] | 56.0 [23 to 77] | 55 [23 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 24 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 21 | 46
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Questionnaire Scale "Intentions for Future Use"
Description: Using the questionnaire scale "Intentions for Future Use" How much each participant intends to use the products in the future.
  Scale: "Think about the product you just used. If this was the only flavor available, how likely would you be to try this flavor again?
  1. Extremely unlikely
  2. Unlikely
  3. Neutral
  4. Likely
  5. Extremely likely The range of observed responses from participants for both groups was 1-5. Not all participants completed all study measures so the number of respondents is lower than enrolled.
Time Frame: during the intervention
Population: Participants who participated in the study
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Tobacco: Participants received a tobacco flavored pod for the electronic cigarette during a 30-minute session with the electronic cigarette. The researcher and participant were blinded to flavor during the visits.
- Menthol: Participants received a menthol-flavored pod for the electronic cigarette during a 30-minute session with the electronic cigarette. The researcher and participant were blinded to flavor during the visits.
Arm/Group | Tobacco | Menthol
Number analyzed (Participants) | 41 | 41
units on a scale | 3.1 [1 to 5] | 3.7 [1 to 5]

2. Secondary Outcome: Questionnaire Scale "Subjective Vaping Experience"
Description: Please indicate how you are feeling right now on a scale from 0 to 100 where 0 is not at all and 100 is extremely.
  How pleasant would the e-cigarette be to use right now? The observed range of responses from participants for both arms was 0 to 100. Not all participants completed all study measures so the number of respondents is lower than enrolled.
Time Frame: during the intervention
Population: Participants who participated in the study
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Tobacco: Participants receive tobacco flavored pod for the electronic cigarette during a 30-minute session with the electronic cigarette. The researcher and participant were blinded to flavor during the visits.
Arm/Group | Tobacco | Menthol
Number analyzed (Participants) | 41 | 41
units on a scale | 38.0 [0 to 100] | 48.1 [0 to 100]

3. Secondary Outcome: Questionnaire Scale "Perceptions of Flavor"
Description: On a scale from 0 to 100 where 0 is not at all and 100 is extremely, to what extent did you like the flavor you just used? The observed range of responses from participants in both arms was from 0 to 100.
  Not all participants completed all study measures so the number of respondents is lower than enrolled.
Time Frame: during the intervention
Population: Participants who participated in the study.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Tobacco | Menthol
Number analyzed (Participants) | 41 | 41
units on a scale | 34.0 [0 to 100] | 51.0 [0 to 100]

4. Secondary Outcome: Questionnaire Scale "Product Demand"
Description: On a scale from 0 to 100 where 0 is not at all and 100 is extremely, how willing would you be to use the flavor you just used again in the future? The observed range of responses from participants in both arms was from 0 to 100.
  Not all participants completed all study measures so the number of respondents is lower than enrolled.
Time Frame: during the intervention
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Tobacco | Menthol
Number analyzed (Participants) | 41 | 41
units on a scale | 38.7 [0 to 100] | 49.7 [0 to 100]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for each participant during the study which ranged from 1 week to 1 month, and were assessed at 6 months after last study visit completion for each participant, a total of up to 7 months.
Description: No different definitions.
Groups:
- Tobacco Pod: Participants receive tobacco flavored pod for the electronic cigarette during the first during the 30-minute session with the electronic cigarette. Then participants received a menthol-flavored pod at the second session. The researcher and participant were blinded to flavor during the visits.
- Menthol Pod: Participants receive menthol flavored pod for the electronic cigarette during the first during the 30-minute session with the electronic cigarette. Then participants received a tobacco-flavored pod at the second session. The researcher and participant were blinded to flavor during the visits.
Arm/Group | Tobacco Pod | Menthol Pod
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT04996940/Prot_SAP_000.pdf